CLINICAL TRIAL: NCT05514522
Title: The UK Interstitial Lung Disease Long-COVID19 Study (UKILD-Long COVID): Understanding the Burden of Interstitial Lung Disease in Long COVID.
Acronym: UKILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); University of Nottingham (Other); University of Southampton (Other); University of Leicester (Other); University of Manchester (Other); University of Liverpool (Other); University of Sheffield (Other); University of Oxford (Other); University College, London (Other); University of Newcastle Upon-Tyne (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 21IC6978
Record Dates: First submitted 2022-08-04; First posted 2022-08-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease; SARS-CoV-2 Infection
Keywords: Interstitial Lung Disease; COVID; PC-ILD population
MeSH Terms: conditions — Lung Diseases, Interstitial; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be taken for plasma/ serum for epithelial and endothelial damage biomarkers, coagulation and genetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study of hospitalised and non-hospitalised patients post- infection with SARS-CoV-2. The study aims to recruit 2000 individuals, with proven COVID-19, who were not hospitalised but presented to Long-COVID clinics with persistent respiratory symptoms such as breathlessness or cough and are referred for cross-sectional imaging (computer tomography, CT) at baseline (3 months weeks after their first COVID-19 symptoms). The study will run for 18 months.

DETAILED DESCRIPTION:
Given the large number of patients infected with SARS-CoV-2, it is vital that the extent of PC-ILD is determined; its natural history defined particularly whether it is time-limited inflammation and reversible, or develops into persistent, or even progressive, fibrosis. Determining the natural history of PC-ILD, and risk factors as well as biomarkers related to outcome such as disease progression, will enable a precise approach to treatments such as immunomodulation or antifibrotic therapy [6], stratification into clinical trials, prognostication and appropriate service provision. This will facilitate assessment and prioritisation of both conventional and novel therapies used in the treatment of COVID-19 during the acute phase to mitigate the subsequent development of PC-ILD. By exploring the long-term implications of SARS-CoV-2 infection across the full spectrum of COVID-19 disease ranging from non-hospitalised patients managed in the community with mild symptoms to those requiring mechanical ventilation, we will define the risk factors for PC-ILD including disease severity, host genetic factors and the effects of antiviral and immunomodulatory treatment administered during the acute phase of the illness. The UKILD Post COVID study is a prospective multicentre observational cohort study that will be managed through the Imperial College National Heart and Lung Institute and funded by the UKRI Medical Research Council and an NIHR professorship (RGJ).

The PHOSP COVID study (ISRCTN10980107) is a national consortium that provides a platform to study the long-term consequences of COVID19 hospitalisations [18]. An expected 10,000 individuals hospitalised by COVID-19 are to be included in baseline assessments after testing positive on PCR for SARS-C0V-2 and will be recruited through the PHOSP platform. The study described here will aim to recruit a further 2000 individuals, with proven COVID-19, who were not hospitalised but presented to Long-COVID clinics with persistent respiratory symptoms such as breathlessness or cough and are referred for cross-sectional imaging (computer tomography, CT) at baseline (3 months weeks after their first COVID-19 symptoms) [19]. A total of up to 12,000 people will be assessed for longitudinal follow up into the UKILD-Post COVID study. Following assessment of Post COVID patients at baseline (~3-6 months post infection as defined above), those with clinical and radiological features suggestive of ILD will be included into the UKILD-Post COVID study population. Where there are contraindications for CT and if clinically indicated, participants will be eligible for a research-guided 3D ultrashort echo time (UTE) proton MRI as a surrogate for CT. Where individuals meet criteria for initial study inclusion (COVID-19 and clinical indication for CT scanning) but have no clinical, radiological or physiological features of ILD they will be invited to enroll as part of the control cohort for follow up.

This protocol details the research partnership between Imperial (BREATHE Respiratory hub partner), and partner organizations.

2 STUDY OBJECTIVES

2.1 Primary objective The primary objective of the study is to determine the prevalence of ILD at 12 months following SARS-CoV-2 infection and whether clinical severity correlates with severity of ILD in survivors.

2.2 Secondary objectives

1. to further define the PC-ILD population, in particular, to describe the emerging phenotypes and risk factors of PC-ILD
2. to determine the natural history of PC-ILD phenotypes longitudinally
3. to explore pathomechanisms of PC-ILD for candidate prognostic and theranostic biomarkers.

2.3 The primary endpoint

1. The primary endpoint of the study is as radiologically confirmed diagnosis of fibrotic or non-fibrotic ILD in the 12 months following COVID-19. Sub-studies will have a co-primary endpoint of change in the radiological extent of PC-ILD.

2.4 The secondary endpoints

1. progressive lung function impairment between 3 and 12 months, defined as ≥10% relative decline in FVC, or ≥10% relative decline in DLco, or increasing radiological extent of PC-ILD using image analysis [20].
2. Resolution of ILD, as defined by ≥10% relative improvement in FVC, DLco, or reduction of radiological extent.
3. Persistence of ILD in those not meeting definition of progression or resolution
4. Presence of interstitial lung abnormalities (ILA) on radiological images that do not meet definition of ILD.
5. A comprehensive series of clinical, molecular, MRI and biochemical parameters will be assessed as biomarkers.

Pre-recruitment evaluations Screening and Eligibility Assessment Patients will be assessed by the clinical teams for eligibility against the inclusion or exclusion criteria.

The clinical teams at the recruiting sites will confirm that patients have been infected with SARS-CoV2 before approaching them. Participants must satisfy all the approved inclusion and exclusion criteria of the protocol. Participants will then be invited to participate and informed consent will be obtained at the start of visit 1. Pre-screening for eligibility will take place prior to consent. It will be done by the direct care team using patient notes. There will be no access to patient identifiable data outside of the direct care team prior to consent.

Screening and eligibility for PHOSP COVID/C-MORE participants For PHOSP-COVID participants, screening and eligibility assessment will occur as per the REC approved protocol (IRAS ID 285439).

All patients can be directed to other relevant post-COVID studies, including but not restricted to POSTCODE and XMAS.

3 STUDY DESIGN Prospective observational study of hospitalised and non-hospitalised patients post- infection with SARS-CoV-2. The study aims to recruit 2000 individuals, with proven COVID-19, who were not hospitalised but presented to Long-COVID clinics with persistent respiratory symptoms such as breathlessness or cough and are referred for cross-sectional imaging (computer tomography, CT) at baseline (3 months weeks after their first COVID-19 symptoms). The study will run for 18 months.

Description of study procedure(s) History and Examination (10 mins) : Medical history, allergies, medications and anthropometric measurements including height, weight, and body mass index will be recorded during the study visit (or taken from the hospital notes. Or PHOPS data)

Blood sample collection (10 mins) :

Samples will be taken for plasma/ serum for epithelial and endothelial damage biomarkers, coagulation and genetics Questionnaires (45 mins) Participants will be provided with seven questionnaires; 36 Short-Form Survey (SF-36), Clinical Frailty Scale (CFS), Patient Health Questionnaire 9 (PHQ9), Montreal Cognition Assessment (MOCA), Dyspnoea-12 score, EQ5D-5L, FACIT-F at the end of each study visit.

There are no investigations required for participants co-enrolled in the PHOSP-COVID study.

3.3 Baseline and follow up assessments Initial patient approach Eligibility assessment by clinical team Study information and invitation letter provided to eligible patients

Visit 1 (~3 months) (Post COVID-19 infection patients)

1. Review of eligibility with participant
2. Obtain written informed consent
3. History and anthropometric measurements, e.g. height, weight, body mass index (BMI)
4. Blood sample (6-10 ml) collection
5. Pulmonary function test (20 minutes)
6. Optional 6-minute walk test (6MWT) (10 minutes)
7. Quality of Life questionnaire (SF-36) (10 minutes)
8. Clinical Frailty Scale (CFS) (5 minutes)
9. Personal health questionnaire (PHQ) (10 minutes)
10. Montreal Cognitive Assessment MOCA (10 minutes)
11. Dyspnea 12 score (10 minutes)
12. EQ5D-5L (10 minutes)
13. FACIT-F questionnaire (10 minutes)

Optional Visit 2 (~6 months) (Post COVID-19 infection patients and matched controls) All visit 1 assessments will be repeated.

Visit 3 (~12 months) (Post COVID-19 infection patients) All visit 1 assessments will be repeated. Visits will be scheduled to take place over 1 day. Visit 2 is optional, Visits 1 and 3 are obligatory.

3.3 Monitoring of clinical events and re-analysis of previous scans (clinically indicated) Clinical outcome data and images from clinical scans for all COVID-19 patients will also be collected from around the time of infection and hospitalisation and follow up. Laboratory analyses and chest imaging results undertaken for clinical reasons will also be collected. Access to participant medical records and any relevant hospital data that is recorded as part of routine standard of care; i.e., CT-Scans, blood results and disease progression data etc. will be obtained with patient consent from hospital electronic patient records and NHS digital

3.4 Sample Handling Blood samples for the analysis of serum inflammatory markers, serum biomarkers of endothelial and epithelial injury and coagulation studies, viral serology, viral PCR, and whole genome sequencing, ribonucleic acid sequencing and flow cytometry in blood will be collected. Analysis of venous blood samples will be performed in local NHS laboratories. If the Participant consents approximately 10 ml of blood will be stored in the Division of Cardiovascular Medicine for further analysis as part of collaborations with other groups. Samples will not be collected from participants who are also participating in PHOSP-COVID

Withdrawal Criteria

Early Discontinuation/Withdrawal of Participants : During the course of the study a participant may choose to withdraw early from the study treatment at any time. This may happen for several reasons, including but not limited to:

* The occurrence of what the participant perceives asintolerable AE.
* Inability to comply with study procedures
* Participant decision

According to the design of the study, participants may have the following three options for withdrawal;

1. Participants may withdraw from active follow-up and further communication but allow the study team to continue to access their medical records and any relevant hospital data that is recorded as part of routine standard of care; i.e., CT-Scans, blood results and disease progression data etc.
2. Participants can withdraw from the study but data and samples obtained up until the point of withdrawal to be retained for use in the study analysis. No further data or samples would be collected after withdrawal.
3. Participants can withdraw completely from the study and withdraw samples collected up until the point of withdrawal. The samples already collected would not be used in the final study analysis.
4. In addition, the Investigator may discontinue a participant from the study at any time if the Investigator considers it necessary for any reason including, but not limited to:

   * Ineligibility (either arising during the study or retrospectively having been overlooked at screening)

Participants that choose to withdraw from the study will not be replaced. The type of withdrawal and reason for withdrawal will be recorded in the CRF. If the participant is withdrawn due to an adverse event, the Investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved or .

ASSESMENT AND FOLLOW UP Optional follow up and assessment

As previously detailed in section 3.3 above, participants will agree to a final follow up assessment and an optional interim assessment

Optional Visit 2 (~6 months) (Post COVID-19 infection patients and matched controls) All visit 1 assessments will be repeated. All visit 1 assessments will be repeated.

Visits will be scheduled to take place over 1 day. Visit 2 is optional, visits 1 and 3 are obligatory. For research specific visits, participants will be offered reimbursement for travel expenses. This includes reimbursement for petrol, car parking, taxis.

Clinical outcome data and images from clinical scans for all COVID-19 patients will also be collected from around the time of infection and hospitalisation and follow up. Laboratory analyses and chest imaging results undertaken for clinical reasons will also be collected. Access to participant medical records and any relevant hospital data that is recorded as part of routine standard of care; i.e., CT-Scans, blood results and disease progression data etc. will be obtained with patient consent from hospital electronic patient records and NHS digital. The end of the study will be the point at which the final patient follow-up and assessment have been completed.

A detailed Image Management protocol for the UKILD-Post COVID Study provides a comprehensive outline of the purpose, operation, methods, policies, and governance of Image collection for UKILD. It describes the procedures used to collect and store images. (appendix 1)

STATISTICS AND DATA ANALYSIS

The prevalence of MDT-confirmed PC-ILD at both early (up to 6 months) and again at late (10-15 month) time-points and will be assessed within the total study population. The prevalence of broader radiological abnormalities and phenotypic patterns will also be assessed in a descriptive analysis, together with demographics, haematological and biochemical profiles, physiological performance, and patient-reported outcome measures. Analyses will be performed overall and stratified according to hospitalised and non-hospitalised, as well as severity of infection in hospitalised patients defined above.

Baseline and longitudinal changes in biomarkers reflecting PC-ILD evolution, including circulating factors and cell-types from detailed serological and cellular analysis, will be assessed in multilevel models for repeated measures to test associations according to the presence or absence of PC-ILD at late time points (10-15 months), and according to progression, resolution, or persistence of radiological patterns over follow up time points.

Analyses will be performed using standard epidemiological and statistical genetics methodology. This will include cross-sectional and longitudinal studies, and analyses of disease prevalence and incidence.

Analysis design and choice of controls will be dependent upon the precise nature of the research question. Identification of risk factors for a specific COVID-19 sequela would involve controls both from within UKILD-Long COVID (without the sequela) and serology-positive controls with prospective questionnaire and healthcare record linkage from Longitudinal Population Studies (for example, UK Biobank, Coronagenes, EXCEED) and pre-existing disease cohorts. Analyses aiming to characterise and understand the clinical features, subtypes and trajectories of sequelae (for example, sarcopaenia) would evaluate the cross-sectional and longitudinal clinical data and biomarkers of UKILD-Long COVID participants who are presenting with the sequelae being studied.

The participant organisations making uo the UKILD-long COVID study group have extensive experience of development of, and collaborative use of, disease-specific and general population cohort studies both nationally and internationally enabling access to control populations and alignment of research strategies for rapid validation and replication of findings.

Statistical significance thresholds will be defined in advance of each analysis and will take into account issues of multiple testing and a priori evidence.

Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

Project statistician: Dr Iain Stewart email:

iain.stewart@imperial.ac.uk National Heart and Lung Institute Guy Scadding Building, Cale Street, London, SW3 6LY

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old -99 years old
2. Evidence of SARS-CoV-2 infection confirmed by PCR or serology 3 months (+/- 6 weeks) earlier
3. Clinical indication for a chest CT scan as per clinician judgment

Exclusion Criteria:

1. Life-limiting illness within 12 months
2. Significant pre-existing lung disease prior to March 2020, which in the investigator's judgement could make the chest CT scans difficult to interpret

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community (Not Hospitalized) participants who have confirmed Evidence of SARS-CoV-2 infection between the age of 18 an 99 with a clinical indication for CT.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Examine and compare the prevalence of ILD in patients with varying severity of COVID-19 | 12 months
  Non-hospitalised will be compared with hospitalised patients and COVID severity defined as varying levels of respiratory support

SECONDARY OUTCOMES:
Determine progressive lung function impairment between 3 and 12 months | 12 months
  >10% relative decline in FVC >10% relative decline in DLco Increasing extent of ILD on CT measured quantitatively Increasing extent of ILD on CT agreed by visual MDT consensus
Resolution of ILD | between 3 and 15 months post-acute SARS-CoV-2
  >10% relative improvement in FVC >10% relative improvement in DLco Decreasing extent of ILD on CT measured quantitatively
Persistence of ILD in those not meeting definition of progression or resolution | between 3 and 15 months post-acute SARS-CoV-2
  Between ±9.9 relative improvement in FVC Between ±9.9 relative improvement in DLco <1% change in extent of ILD on CT measured quantitatively
Breathlessness | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Statistically significant differences between groups for patient reported measures using one or more of the following validated questionnaires:
  Medical Research Council dyspnoea scale (breathlessness) Dyspnoea 12 (breathlessness) FACIT-F (fatigue) Montreal Cognition Assessment (MOCA)
Measure quality of life | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Statistically significant differences between groups for patient reported measures of quality of life using one or more of the following validated questionnaires:
  Short Form -36 (SF-36) EQ5D-5L
impact of COVID19 on aerobic capacity and endurance | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Statistically significant differences between groups for physical tests including one or more of the following:
  Incremental shuttle walk test Cardiopulmonary exercise test
Exploratory biomarkers correlated with ILA/ILD | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Statistically significant differences in circulating biomarkers as measured using one of more of the following:
  Whole blood RNA sequencing Peripheral blood mononuclear cell single cell RNA sequencing
Compare serological and cellular measures of epithelial and endothelial injury and thrombosis | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Serum biomarkers of epithelial and endothelial injury, NETosis and thrombosis Cellular measurements in these same patients. Serum/ Plasma: Nordic biomarkers, LRG-1, MMP-7 etc; NETs
Compare genetic risk factors for lung fibrosis and radiological progression, continuously and dichotomised | No sooner than 3 month visit
  genome-wide array genotyping Genetic testing from blood/ saliva of putative candidate genes and use of GENOMIC data, and telomere length in a subset
Assess the relationship between routinely collected laboratory parameters markers | 3 month, 6 months (+/- 6 weeks) and 12 months (+/- 3 months) post SARS-CoV-2 infection
  Statistically significant differences in routinely-collected blood and urine measures including:
  CRP FBC

CONTACTS AND LOCATIONS:
Overall Officials: Gisl Jenkins, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Final results of the study will be disseminated in the form of a manuscript/s in a peer-reviewed journal scientific journals, presented at national and international conferences and in local meetings. In addition, where relevant, data from potential interim analyses will be presented at (a) relevant congress (es). In addition, the study database will be made available for future research.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05514522/Prot_SAP_001.pdf